CLINICAL TRIAL: NCT05976113
Title: Multiple Classifier Endometrial Cancer
Brief Title: A Retrospective Study on Multiple Classifier Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 1402020
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multiple classifier endometrial cancer: Endometrial cancer patients who have two or more molecular features
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — Just obsrevation following standard of care (including surgery, chemotherapy and radiation when appropriate)

SUMMARY:
Endometrial cancer is not a single entity but rather a very heterogeneous group of diseases. Historically, endometrial cancer patients have been classified as endometrioid (type I) or non-endometrioid (type II) according to the dualistic Bokhman model- However, this approach has been limited in accurately predicting prognosis and guiding treatment owing to heterogeneity within subtypes, inadequate incorporation of molecular and genetic information, and high interobserver variability .

In the last ten years, after the publication of The Cancer Genome Atlas (TCGA)[5], the molecular classification of endometrial cancer into four molecular subtypes [(i) POLE/ultramutated group (POLE mutated), (ii) mismatch repair deficiency/microsatellite-instable, hypermutated group (MMRd/MSI-H), (iii) copy-number-high, TP53-mutant (CNH/p53abn), and (iv) copy-number-low, TP53-wild-type (CNL, or No Specific Mutational Profile [NSMP])] has rapidly gained interest. Recently, the European Societies of Gynaecological Oncology, Radiotherapy and Oncology, and Pathology (ESGO-ESTRO-ESP), the European Society of Medical Oncology (ESMO), the National Comprehensive Cancer Network (NCCN), and the new 2023 International Federation of Gynecology and Obstetrics (FIGO) staging system have promoted the use of (surrogate) molecular classification. Retrospective studies supported the value of adopting molecular classification to offer reliable data on prognostication and adjuvant treatment decisions. Although no prospective data are available, current guidelines promote the use of molecular profiles to tailor adjuvant treatment after surgery. As only a few retrospective studies have investigated the association between molecular profiles and response to various adjuvant treatments, it is important to note that data are limited. Interestingly, the growing adoption of molecular profiling led to the detection of a subgroup of tumors called multiple classifiers, characterized by multiple (two or three) molecular features. According to the guidelines, tumors with a POLE mutation should be considered POLEmut, regardless of other molecular features, whereas MMRd/MSI-H tumors with a p53 abnormality should be considered MMRd/MSI-H. Data on these patients is limited and fragmentary. The aforementioned consensus is based solely on a large retrospective cohort of multiple classifiers collected by Leon-Castillo et al.. Hence, to fill this literature gap, the investigators designed this retrospective study, which aimed to collect multiple classifiers patients to improve knowledge on this emerging category.

ELIGIBILITY:
Inclusion criteria were the following: (i) histological diagnosis of endometrial cancer; (ii) execution of hysterectomy (with or without salpingo-oophorectomy) with or without nodal dissection; (iii) apparent early-stage disease; (iv) conventional pathological evaluation; and (v) molecular/genomic evaluation of the disease (including at least POLE sequencing, MMR protein immunostaining or MSI assessment, p53 immunostaining or TP53 sequencing). Exclusion criteria were: (i) consent withdrawal, (ii) execution of neoadjuvant therapy, and (iii) stage IV disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients with uterine cancers
Study Population: This is a retrospective study with patients diagnosed with multiple classifier endometrial cancer Data of consecutive patients treated between June 1, 2019, and January 31, 2023, were collected.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided